# Personalizing intervention to reduce clinical inertia in the treatment of hypertension

Principal Investigator: Nancy Haff, MD, MPH

Identifier: NCT04603560

Consent form date: September 28, 2021

# **CONSENT PROCESS**

Physician subjects will be invited to participate via email. The information sheet below will be attached to the email, and contains information about the study, their participation, and the names and contact information for study staff who can be reached for a phone or video conversation if they have any questions or concerns.

Interested physicians will be asked to click on a link in the email to open a secure RedCap survey. There, physicians will again view an electronic copy of this information sheet. If the physician agrees to participate, he or she will click a button indicating "I agree".

#### HYPERTENSION STUDY INFORMATION SHEET

#### Overview

This is a study about the treatment of hypertension in primary care. We are specifically interested in how to help primary care physicians and patients achieve blood pressure goals.

We are asking you to take part in this study because you are a primary care physician at Massachusetts General Hospital (MGH) who treats patients with hypertension. About 45 primary care physicians at MGH will participate in the study.

#### **Participation**

If you decide to join this research study, the following things will happen:

- 1) We will ask you to complete an **online survey** designed to measure personality traits and behavioral tendencies. The survey is expected to take **10-15 minutes**.
- 2) You will then be randomly assigned to one of three study groups. One group will receive once-weekly emails with information about their patients with hypertension. Another group will receive an average of 1-2 inbasket messages per week about their patients with hypertension. The third group will not receive any messages. It is always your choice whether or not to act on the information that you receive. This portion of the study will last approximately 3-4 months.
- 3) You may be invited to participate in a virtual, structured interview via an MGB-approved video platform at the end of the study to discuss barriers and facilitators of hypertension treatment. Only some providers will be asked to participate. We expect each interview to last 30-45 minutes.
- 4) The remainder of the data for the study will be collected using routinely documented information in Epic and will not require any additional documentation or effort on your part.

#### Risks, Benefits, and Privacy

We expect there to be minimal risks to participating in this study.

The EHR in-basket/email support designed for this trial is meant to highlight guideline-based information that could be useful for hypertension management and prescribing. The primary risk of participation is breach of confidentiality.

To protect privacy, surveys will be completed using REDCap, a secure, HIPPA compliant webbased application. Data will only be identifiable to the MGB researchers with access to a password-protected, REDCap database.

If you are invited to participate in a follow-up interview, we will audio-record virtual interviews but will not record any identifiable information about you, and we will safeguard those recordings. Your participation is voluntary, and you can decline or stop at any time. We will request your permission for the collection of audio recordings from the interview.

Efforts will be made to limit the use and disclosure of your personal information, including research study records, to people who have a need to review this information. We cannot promise complete secrecy. Organizations that may inspect and copy your information include the IRB and other representatives of this institution.

You should not expect to gain any direct benefit from taking part in this study. We hope patients in need of treatment intensification for hypertension will benefit in the future from this research.

Your participation is voluntarily, and you can stop at any time. If you choose not to participate in this study at any point, it will not affect your professional standing or evaluations with the department.

### **Payment**

You will be paid for participation in this study: \$75 for the baseline questionnaires, and an additional \$100 if you are invited and complete a post-study interview. This remuneration will be provided by check. To process the checks, study staff will need your name, address, and SSN. You will have the option to provide this via the HIPAA-secure REDCap survey or over the phone directly to a study staff member at your convenience. This information will only be used for payment purposes and will be destroyed after payments are complete.

## **Study Title and Sponsor:**

<u>Title: Personalizing intervention to reduce clinical inertia in the treatment of hypertension</u> Sponsor: National Institute on Aging.

## **Study Contacts**

Research Assistant: Katie Crum

Phone: 617-264-3094

Email: kcrum1@bwh.harvard.edu

• Principal Investigators: Nancy Haff, MD, MPH

Phone: 857-307-3826 Email: <a href="mailto:nhaff@partners.org">nhaff@partners.org</a>

Niteesh Choudhry, MD, PhD

Phone: 617-278-0930

Email: nchoudhry@bwh.harvard.edu

Please reach out to any of contacts above if you have any questions or concerns at any time.

If you'd like to speak to someone not involved in this research about your rights as a research subject, or any concerns or complaints you may have about the research, contact the Partners Human Research Committee at 857-282-1900.